CLINICAL TRIAL: NCT06659055
Title: Bone Mineral Density Assessment Using Dual-energy Stereoradiography: Agreement Between BMD T-scores From EOSedge™ Versus Traditional DXA - BMD Agreement Study
Brief Title: Bone Mineral Density Agreement Study Between EOSedge™ Versus Traditional DXA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ATEC.EOS-2402
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Indicated for EOSedge Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Volunteers (Other): Healthy volunteers will undergo EOSedge and DXA imaging
  Interventions: Radiation: DXA Imaging; Radiation: EOSedge imaging
- Subjects indicated for EOSedge imaging (Other): Subject receiving EOSedge imaging as SOC will also receive an additional DXA scan.
  Interventions: Radiation: DXA Imaging

INTERVENTIONS:
Radiation: DXA Imaging — DXA imaging: lumbar spine, bi-lateral femoral necks
Radiation: EOSedge imaging — Full body or full spine image
  Arms: Healthy Volunteers

SUMMARY:
The purpose of this research is to collect medical imaging data to allow for the comparison of bone mineral density measurements from two different types of low-dose x-ray exams, EOSedge and conventional DXA. The main question it aims to answer is:

Is there agreement between the calculated T-scores between the 2 different types of x-ray exams?

DETAILED DESCRIPTION:
This is a multi-center, prospective, controlled, cross-sectional agreement study of subjects indicated for radiography using EOSedge biplanar full-body or full-spine imaging OR volunteers undergoing non-diagnostic imaging.

From the potential pool of EOSedge examinees, screening data will be reviewed to determine further eligibility. Subjects who sign an informed consent form and meet all inclusion criteria and none of the exclusion criteria will be asked to participate in the study.

Subjects who consent to participate will be enrolled from the time of consent through completion of evaluable image acquisition which will include both EOSedge and DXA scans.

EOSedge exams will be performed as is typical for the evaluation of spinal and/or other orthopaedic conditions, and the output will be collected for post-hoc computation of BMD.

DXA exams will be study-prescribed (or standard of care if consistent with this protocol) and ideally performed on the same day as EOSedge exams (but may be scheduled as much as 60 days apart).

In addition to the radiographic imaging from which spinal/postural alignment parameters may be obtained, some demographic and diagnostic details about the subject will be captured via study-specific case report forms (CRFs). Subjects will also complete a questionnaire that every subject fills out prior to having a DXA scan according to ISCD guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Observational Arm:

   o Subjects at clinical sites, indicated for full-spine or whole-body radiography via EOSedge 2E biplanar imaging (e.g., in the preoperative evaluation of spine and/or other orthopaedic conditions) as part of their routine medical care. Participants may already have completed their routine imagining, or may be scheduled to undergo it within 60 days of study enrollment.
2. Interventional Arm:

   o Volunteers at non-clinical sites, who meet the criteria to undergo non-diagnostic imaging, as part of a research study.
3. Male or female subjects who are at least 20 years of age at the time of imaging acquisition
4. Written informed consent obtained from the potential subject and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

1. Subjects who have been administered contrast agents or radionuclides within 7 days prior to scheduled radiographic imaging (EOS and DXA)
2. Subjects who are pregnant or wanting to become pregnant during the timeframe of study participation (due to risks associated with radiographic imaging)
3. Subjects with a BMI ≥ 35 kg/m2
4. Subjects known to have severe degenerative changes or fracture deformity in the measurement area (i.e., lumbar spine L1-L4, bilateral femoral neck/trochanter; note that unilateral femoral evaluation is acceptable), as defined by the Investigator's determination of the likelihood of reasonably assessing bone mineral density of those areas
5. Subjects known to have implants, hardware, devices, or other foreign material in the measurement area (i.e., lumbar spine L1-L4, bilateral femoral neck/trochanter; note that unilateral femoral evaluation is acceptable)
6. Subjects unable to attain correct position and/or remain motionless for the measurement (e.g., subjects unable to stand unassisted in the EOS unit, or to lie appropriately in the DXA scanner)
7. Subjects known to have extra or missing lumbar vertebrae (i.e., more or fewer than 5 mobile lumbar segments)
8. Subjects participating in another clinical study which may compromise this study's results or compliance with this study's procedures
9. Subjects with presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
AP Spine T-score Agreement | between 0-60 days
  Calculation of EOSedge BMD will be post-processed from the bi-planar EOSedge 2E radiographs, and is measured in g/cm² surface mass on four lumbar vertebrae (L1-L4) in the anteroposterior (AP) projection. BMD results from the conventional DXA system will be similarly acquired from the spine (AP L1-L4) exam, and the paired T-scores derived from the BMD results will be tested for statistical agreement across the two systems.

SECONDARY OUTCOMES:
Hip T-score Agreement | between 0-60 days
  Calculation of EOSedge BMD will be post-processed from the bi-planar EOSedge 2E radiographs, and is measured in g/cm² surface mass at the femoral neck in the anteroposterior (AP) projection. BMD results from the conventional DXA system will be similarly acquired from the hip exam, and the paired T-scores derived from the BMD results will be tested for statistical agreement across the two systems.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Honor Health, Phoenix, Arizona
  - ATEC Carlsbad, Carlsbad, California
  - ATEC Mephis, Memphis, Tennessee
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided